CLINICAL TRIAL: NCT06687057
Title: A Heart Rate Variability (HRV) Biofeedback Training to Reduce Symptomatology Associated With Functional Gastrointestinal Disorders (FGID) in College Students.
Brief Title: A Heart Rate Variability (HRV) Biofeedback Training in Functional Gastrointestinal Disorders (FGID)
Acronym: BF_FDGI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Collaborators: University of Padova (Other); Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Eleonora Volpato, Principal Investigator, Fondazione Don Carlo Gnocchi Onlus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UCSC_123_24
Record Dates: First submitted 2024-11-10; First posted 2024-11-13 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Functional Gastrointestinal Disorders (FGIDs)
MeSH Terms: conditions — Gastrointestinal Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biofeedback (Experimental): The actual administration of the HRV-Biofeedback protocol: 5 HRV biofeedback training sessions of 45 minutes each, conducted biweekly.
  Interventions: Behavioral: HRV Biofeedback Training
- Placebo (Placebo Comparator): Placebo condition: 5 control sessions of 45 minutes each, conducted biweekly.
  Interventions: Other: Placebo Training

INTERVENTIONS:
Behavioral: HRV Biofeedback Training — The intervention involves 5 training sessions lasting 45 minutes (specifically, 5-minute baseline and 5 HRV biofeedback trials lasting 5 minutes each) according to the protocol published by Lehrer et al. (2013). Physiological signals (ECG and respiratory rate) will be recorded during all sessions. During the training, participants will see on the screen a graph representing heart rate superimposed on a graph representing abdominal breathing. They will be asked to synchronize the two signals so that the changes in heart rate are in phase with the respiratory cycle in order to maximize the difference between the maximum and minimum heart rate within each respiratory cycle [i.e., respiratory sinus arrhythmia (RSA), an index of vagal modulation on the heart] (Lehrer et al., 2003; Lehrer et al., 2000).
  Arms: Biofeedback
Other: Placebo Training — The Placebo procedure requires participants to attend 5 sessions lasting 45 minutes during which they perform a task. Physiological signals (ECG and respiration rate) will be recorded during all sessions. Participants will see on the screen a graph representing heart rate superimposed on a graph representing abdominal breathing but these will not directly reflect the subject's cardiorespiratory activity. Participants in the control group will be asked to synchronize the two signals so that the changes in heart rate are in phase with the respiratory cycle, but the feedback on the screen will not reflect that subject's RSA changes.
  Arms: Placebo

SUMMARY:
Functional Gastrointestinal Disorders (FGIDs) are conditions characterized by chronic gastrointestinal symptoms without evidence of pathology. These disorders are believed to result from alterations in gut-brain communication. The most common subtypes are Irritable Bowel Syndrome (IBS) and Functional Dyspepsia (FD), often accompanied by chronic pain, anxiety, and depression. The role of stress in the manifestation of FGIDs is notable, with stress-related distress affecting the nerve pathways that connect gut and brain. Recent interest has focused on the use of Heart Rate Biofeedback (HRV). High levels of stress are associated with reduced HRV, which is common in patients with FGID. HRV biofeedback has been shown to be effective in improving parasympathetic tone and reducing sympathetic tone. The present study aims to evaluate the effectiveness of this approach in reducing stress and symptoms associated with FGIDs in college students.

The project involves online screening to recruit participants, who will then be randomized to receive either the true HRV biofeedback treatment or a placebo condition. Pre- and post-treatment assessments include psychological questionnaires, physiological recordings, and a three-month follow-up. The treatment is expected to improve HRV, thereby reducing anxiety and gastrointestinal symptoms.

ELIGIBILITY:
Inclusion Criteria:

* presence of clinically significant anxiety symptoms (DASS-21 > 4)
* presence of symptoms related to Functional Gastrointestinal Disorders (in English, known as Functional Gastrointestinal Disorders (FGIDs)) (IBS-SSS > 75);
* obtaining informed consent to participate in the study;
* Absence of organic gastrointestinal diseases: thus, they will be excluded if with a current or previous diagnosis of intestinal disease (e.g., ulcerative colitis);
* absence of clinical conditions including neurological disorders (previous head trauma, degenerative neurological disorders, stroke, etc.) and cardiovascular disorders (hypertension, cardiac arrhythmias, etc.).

Exclusion Criteria:

* absence of clinically significant anxiety symptoms (DASS-21< 4);
* absence of symptoms related to Functional Gastrointestinal Disorders (in English, known as Functional Gastrointestinal Disorders (FGIDs)) (IBS-SSS < 75);
* lack of obtaining Informed Consent to participate in the study;
* presence of organic gastrointestinal diseases: therefore, they will be excluded if with a current or previous diagnosis of intestinal disease (e.g., ulcerative colitis).
* presence of clinical conditions including neurological disorders (previous head trauma, degenerative neurological disorders, stroke, etc.) and cardiovascular disorders (hypertension, cardiac arrhythmias, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Anxiety | Day 0 (T0); Week 4 (T1); Month 3 (T2)
  The Depression Anxiety Stress Scales - 21 (DASS-21) is 21-item self-report measure designed to assess the severity of general psychological distress and symptoms related to depression, anxiety, and stress in adults older adolescents (17 years +).
Stress | Day 0 (T0); Week 4 (T1); Month 3 (T2)
  The Depression Anxiety Stress Scales - 21 (DASS-21) is 21-item self-report measure designed to assess the severity of general psychological distress and symptoms related to depression, anxiety, and stress in adults older adolescents (17 years +).
Emotion Regulation | Day 0 (T0); Week 4 (T1); Month 3 (T2)
  The Emotion Regulation Questionnaire (ERQ) is composed of ten items divided into two factors: cognitive reappraisal with six items and expressive suppression with four items. It is answered on a Likert scale ranging from 1 (total disagreement) to 7 (total agreement).
Irritable Bowel Severity | Day 0 (T0); Week 4 (T1); Month 3 (T2)
  This scale evaluates primarily the intensity of IBS symptoms during a 10-day period: abdominal pain, distension, stool frequency and consist- ency, and interference with life in general. The IBS-SSS calculates the sum of these 5 items each scored on a visual analog scale from 0 to 100. Although the IBS-SSS uses patient-rated intensity of IBS symptoms, the determination of severity by the scoring system was originally anchored to a physician's assessment of patient severity.
Heart Rate Variability | Day 0 (T0); Week 4 (T1); Month 3 (T2)
  Electrocardiogram (ECG) and Heart Rate Variability in particular, recorded through three Ag/AgCl electrodes placed with a proximal type fitting, using the second Einthoven lead. Heart rate and HRV parameters in time and frequency and nonlinear indices will be extracted from the ECG. They will also be monitored during the proposed training (experimental and control).

SECONDARY OUTCOMES:
Interception | Day 0 (T0); Week 4 (T1); Month 3 (T2)
  The Body Perception Questionnaire (BPQ) is a self-report measure of body awareness and autonomic symptoms (i.e. symptoms experienced in organs innervated by the ANS). Its items are based on the organization of the autonomic nervous system (ANS), a set of neural pathways connecting the brain and body.
Emotional State | Day 0 (T0); Week 4 (T1); Month 3 (T2)
  The PANAS is a self-report measure used to assess levels of positive and negative affect. It consists of 20 items asking the extent to which the respondent has experienced different emotions during a given timeframe.
Respiratory Rate | Day 0 (T0); Week 4 (T1); Month 3 (T2)
  Respiratory rate (RR) recorded through bands (strain gauges) placed around the chest and around the abdomen. It will be monitored during both the experimental and control treatments
Depression | Day 0 (T0); Week 4 (T1); Month 3 (T2)
  The Depression Anxiety Stress Scales - 21 (DASS-21) is 21-item self-report measure designed to assess the severity of general psychological distress and symptoms related to depression, anxiety, and stress in adults older adolescents (17 years +).

CONTACTS AND LOCATIONS:
Locations (1):
- Eleonora Volpato, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Lehrer PM, Vaschillo E, Vaschillo B, Lu SE, Eckberg DL, Edelberg R, Shih WJ, Lin Y, Kuusela TA, Tahvanainen KU, Hamer RM. Heart rate variability biofeedback increases baroreflex gain and peak expiratory flow. Psychosom Med. 2003 Sep-Oct;65(5):796-805. doi: 10.1097/01.psy.0000089200.81962.19. PMID 14508023
- [Result] Mather M, Thayer J. How heart rate variability affects emotion regulation brain networks. Curr Opin Behav Sci. 2018 Feb;19:98-104. doi: 10.1016/j.cobeha.2017.12.017. PMID 29333483
- [Result] Goessl VC, Curtiss JE, Hofmann SG. The effect of heart rate variability biofeedback training on stress and anxiety: a meta-analysis. Psychol Med. 2017 Nov;47(15):2578-2586. doi: 10.1017/S0033291717001003. Epub 2017 May 8. PMID 28478782